CLINICAL TRIAL: NCT00948948
Title: Mentor Adjunct Study for Silicone Gel-Filled Mammary Prosthesis
Acronym: Adjunct
Status: Approved for marketing | Type: Expanded Access
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0005033; NCT00495937 (obsolete NCT alias); NCT00582153 (obsolete NCT alias)
Record Dates: First submitted 2009-07-08; First posted 2009-07-29 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Breast Reconstruction

INTERVENTIONS:
Device: Silicone Gel-Filled Mammary Prostheses — Mentor Gel-Filled Mammary Prostheses are comprised of a shell made of medical grade silicone elastomer. Gel-filled implant devices manufactured by Mentor will be used in this study:
  * Gel-filled device which is available in smooth surface and textured surface (Siltex®)
  * Becker Expander/Mammary Prosthesis which is available in both the smooth and the textured (Siltex) version
  Both of these devices were originally indicated for both augmentation and reconstruction mammaplasty procedures, however for purposes of this study, indications are for reconstruction only.

SUMMARY:
Mentor is undertaking a five-year prospective clinical study designed to collect safety data associated with the implantation of its gel-filled mammary prostheses. This study is an "adjunct" study, which will encompass clinical reviews of reconstructive cases in all patients who meet clinical and regulatory criteria for breast reconstruction with gel-filled mammary prostheses. This "adjunct" study will be accomplished under a limited clinical protocol in which specific parameters will be required but with controls somewhat less stringent than those normally required in Investigational Device Exemption (IDE) Trials.

DETAILED DESCRIPTION:
Objectives of this study are to gather safety data regarding short term, post-implant events and complications needed to support Premarket Approval (PMA) submissions for Mentor Silicone Gel-Filled Mammary Prostheses and to maintain a comprehensive record of the patient's ongoing medical history. The FDA has placed the devices in a regulatory category as a Class III device, pursuant to the Medical Device Amendments to the Federal Food and Drug Act which went into effect in May 1976. For devices in this class, FDA requires certain clinical data regarding the risks associated with mammary prostheses. Due to several issues surrounding possible risks of silicone gel-filled breast implants, the FDA has mandated specific clinical study requirements to further assess possible risks and complications of silicone devices. Clinical data collected via this study will supplement data which will be collected in more extensive "Core" studies for breast reconstruction and augmentation procedures.

Primary Objective - Safety Assessment

Specifically, data collected during this study will provide risk and complication data with regard to short-term use of silicone breast implants. This safety assessment will include, but is not limited to:

* Incidence of capsular contracture
* Occurrence of complications such as infection and seroma
* Rupture rates for the implant

Secondary Objectives

This study is not intended to assess rare, long-term or speculative conditions which are not proven clinically to be associated with mammary prostheses, such as their relationship to Connective Tissue Disorders, an increased risk of cancer or teratogenic effects among breast implant patients. This study is also not intended to address issues regarding the effects of breast implants on mammography interpretation and occurrence of calcium deposits in the tissue surrounding the implant. However, data on these and other complications noted in this study, should they occur, will be recorded and analyzed with regard to the objective of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be female (genotypical females only), and
2. The patient must be willing to follow the study requirements to include:

   1. Sign the Informed Consent Document before surgery is performed. (If the patient is under the age of consent, the parent or guardian must sign. It is the responsibility of the doctor to determine the state's age of majority.)
   2. Agree to complete all required follow-up visits.
   3. For those patients who wish to participate in the Patient Registry: agree to conditions of the Implant Registry and follow the requirements of the Registry program.
   4. Agree to follow Mentor Standard Operating Procedures for explant analysis in which case the patient may be asked to authorize the sponsor to complete analysis on any study device(s) that may require removal throughout the duration of the study.
   5. Must be determined by the Investigator and other medical specialists (as required) to be an acceptable candidate for reconstructive breast surgery. General medical condition and history, as well as psychological appropriateness should be considered before surgical intervention, AND
3. In the medical opinion of the surgeon conditions must be such that saline implants are deemed unsuitable for the patient. (Patient preference for gel implants is NOT considered a medical condition.) Examples of saline unsuitability are:

   1. Severe wrinkling of an existing saline implant to the extent that it would be considered a severe deformity (implant must have been in place longer than 6 months)
   2. Unilateral replacement (opposite breast is gel)
   3. Tissue or skin is too thin to support a saline implant
   4. Previously dissected pocket is incompatible with saline implant, AND
4. The patient must have one or more of the following breast conditions:

   1. Post-unilateral or bilateral mastectomy (immediate or delayed) as a result of cancer or other disease process.
   2. Require reconstruction due to cancer treatments other than mastectomy.
   3. Require a revision due to complications or other undesirable results of a previous surgery for the above reasons.
   4. Post-Trauma defined as total or partial removal of the breast(s) through surgery (for any reason) or as a result of the trauma itself.
   5. Congenital deformities defined as:

      * Pectus Excavatum defined as congenital concave chest wall deformity with abnormalities of the sternum and anterior ribs.
      * Pectus Carinatum defined as convex chest wall deformity with abnormalities of the sternum and anterior ribs.
      * Severe asymmetry defined as congenital or acquired substantial discrepancy in breast sizes such as to represent a significant physical deformity or abnormality (e.g., Poland's syndrome).
   6. Severe ptosis defined as requiring a reconstruction procedure such as a mastopexy (tissue and/or skin must be removed from the breast to qualify as a mastopexy procedure).
   7. Patients who require revision with implant replacement for severe deformity caused by medical or surgical complications, regardless of original indication for implantation or type of device originally implanted.
   8. Replacement or revision for patients whose prior surgery was not a result of treatment for cancer and for whom saline implants are unsuitable (e.g., skin too thin, insufficient tissue, etc.) as deemed by the surgeon.
   9. Size changes (larger or smaller) are only allowed if the Investigator determines that a revision or replacement is required for medical reasons. In a case where a change of size is the only indication for surgery, and no medical necessity exists, the protocol will not allow replacement.
   10. Patients who require Augmentation mammaplasty in the unaffected breast as a result of the surgery, due to one of the above indications, in the affected breast (i.e., unilateral mastectomy with augmentation to opposite breast to provide symmetry).
   11. Special circumstances for implantation will be considered on a case by case basis per written FDA authorization.

Exclusion Criteria:

In addition to general conditions which, in the opinion of the surgeon and/or consulting physicians may exclude a patient from enrollment as a study subject, patients must be excluded if they meet any one of the following conditions.

1. Augmentation mammaplasty and the failure to have at least one of the diagnoses identified in the inclusion criteria.
2. Have an abscess or infection anywhere in their body at the time of study entry.
3. Be currently pregnant or nursing.
4. Be diagnosed as having lupus defined as Systemic Lupus Erythematosus or Discoid Lupus, or scleroderma defined as Progressive Systemic Sclerosis.
5. Currently have uncontrolled diabetes or any diseases which are clinically known to impact wound healing ability.
6. Demonstrate tissue characteristics which are clinically incompatible with mammaplasty (e.g., tissue damage resulting from radiation, inadequate tissue, compromised vascularity or ulceration).
7. Possess any condition or currently be under treatment for any condition, which in the opinion of the Investigator and/or consulting physician(s), may constitute an unwarranted surgical risk.
8. Demonstrate psychological characteristics such as inappropriate attitude or motivation, which, in the opinion of the Investigator are incompatible with the risks, involved with the surgical procedure and the prosthesis.
9. Unwillingness to undergo any further surgery for revision (if required).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sue Schwefel, Study Director — Mentor Worldwide, LLC
Locations (1):
- Mentor Worldwide LLC, Santa Barbara, California, United States